CLINICAL TRIAL: NCT05995392
Title: A Single-Center, Prospective Randomized, Double-Masked, Placebo-Controlled, Parallel- Group Pilot Study of the Effects and Safety of Topical Spironolactone Ophthalmic Solution, 0.005 mg/cc in Subjects With Dry Eye
Brief Title: The Effects and Safety of Topical Spironolactone Ophthalmic Solution, 0.005 mg/cc in Subjects With Dry Eye Disease
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Richard W Yee, MD (Other)
Responsible Party: Sponsor-Investigator, Richard W Yee, MD, Sponsor-Investigator, Yee, Richard W., M.D.
Organization: Yee, Richard W., M.D. (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S2023
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment (Experimental): Subjects receive topical spironolactone ophthalmic solution, 0.005 mg/cc four times a day for 4 weeks.
  Interventions: Drug: Topical spironolactone ophthalmic solution, 0.005 mg/cc
- Placebo (Placebo Comparator): Subjects receive topical spironolactone vehicle as placebo four times a day for 4 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topical spironolactone ophthalmic solution, 0.005 mg/cc — Used four times a day in both eyes for 4 weeks.
  Arms: Treatment
Drug: Placebo — Used four times a day in both eyes for 4 weeks.
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the clinical efficacy of topical spironolactone ophthalmic solution, 0.005 mg/cc in subjects with dry eye disease compared to placebo. The hypothesis for this study is that topical spironolactone ophthalmic solution will be beneficial in the management of signs and symptoms of dry eye disease when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* SANDE questionnaire ≥30 mm
* Schirmer test without anesthesia ≥2 mm/5 minutes
* Corneal fluorescein staining score of ≥1 (0-3 point scale) in at least 1 corneal region of the 5 zones based on the NEI scale, with particular attention paid to the inferior region
* The same eye (eligible eye) must fulfill all the above criteria
* No lagophthalmos, entropion, ectropion
* No significant conjunctivochalasis (graded <2 on a 0-4 point scale)
* Best corrected distance visual acuity (BCDVA) score of +0.7 or better as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) (20/200 Snellen value) in both eyes at the baseline visit
* Intraocular pressure of ≥10 to <21 mmHg
* If a female of childbearing potential, have a negative pregnancy test
* Only patients who satisfy all Informed Consent requirements may be included in the study
* The patient must read, sign and date the Informed Consent document before any study related procedures are performed
* The Informed Consent form signed by patients must have been approved by the Institutional Review Board (IRB) / Independent Ethics Committee (IEC) for the current study
* Patients must have the ability and willingness to comply with study procedures
* Ability to speak and understand the English language sufficiently to understand the nature of the study, to provide written informed consent, and to allow the completion of all study assessments

Exclusion Criteria:

* Evidence of an active ocular infection, in either eye
* Presence of any other ocular disorder or condition requiring topical medication during the entire duration of study
* History of severe systemic allergy or of ocular allergy (including seasonal conjunctivitis) or chronic conjunctivitis and/or keratitis other than dry eye
* Intraocular inflammation defined as Tyndall score >0
* Systemic disease not stabilized within 1 month before Visit 1 (e.g. diabetes with glycemia out of range, thyroid malfunction) or judged by the investigator to be incompatible with the study (e.g. current systemic infections) or incompatible with the frequent assessment required by the study
* Patient had a serious adverse reaction or significant hypersensitivity to any drug or chemically related compounds or had a clinically significant allergy to drugs, foods, amide local anesthetics, or other materials including commercial artificial tears that is judged by the investigator to be incompatible with the study
* Females of childbearing potential (those who are not surgically sterilized or post- menopausal for at least 1 year) are excluded from participation in the study if they meet any one of the following conditions:

  1. are currently pregnant
  2. have a positive result at the urine pregnancy test (Baseline/Day 0)
  3. intend to become pregnant during the study treatment period
  4. are breast-feeding
  5. are not willing to use highly effective birth control measures, such as: hormonal contraceptives - oral, implanted, transdermal, or injected - and/or mechanical barrier methods - spermicide in conjunction with a barrier such as a condom or diaphragm or Intra Uterine Device (IUD) - during the entire course of and 30 days after the study treatment period ends
* Any concurrent medical condition, that in the judgment of the PI, might interfere with the conduct of the study, confound the interpretation of the study results, or endanger the patient's well-being
* Use of topical, nasal, or oral antihistamine within 24 hours prior to or during study enrollment
* Use of oral spironolactone within 6 months prior to or during study enrollment
* Previous use of topical spironolactone ophthalmic solution
* Unstable use of topical cyclosporine, topical corticosteroids, artificial tears, lid scrubs, or any other topical drug for the treatment of dry eye in either eye prior to and during study enrollment
* Contact lenses use at any time 30 days prior or during study enrollment
* Cauterization of the punctum or punctal plugs placed within 14 days prior or during study enrollment
* Any prior ocular surgery (including refractive palpebral and cataract surgery) within 90 days of study enrollment
* History of drug addiction or alcohol abuse
* Participation in a trial with a new active substance during the past 6 months
* Participation in another trial study at the same time as the present study
* Have been exposed to any investigational drug within the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 4 in the Symptom Assessment Questionnaire Dry Eye (SANDE) score. | Baseline to Week 4
  The SANDE score is calculated by taking the square root of the product of the severity of symptoms score and the frequency of symptoms score. The SANDE scale ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms and 0 being the minimal amount or absence of dry eye symptoms.

SECONDARY OUTCOMES:
Change from Baseline to Week 4 in the corneal fluorescein staining | Baseline to Week 4
  Corneal fluorescein staining is measured by the 0-3 point National Eye Institute (NEI) grading scale in any one corneal region. 0 represents no staining and 3 represents maximal/severe staining and damages to the cornea. Scores from each of the five corneal regions as defined by the NEI grading scale will be evaluated independently.

OTHER OUTCOMES:
Change from Baseline to Week 4 in SANDE severity sub-score (0-100 point VAS) | Baseline to Week 4
  The SANDE severity sub-score ranges from 0 to 100 with 100 being the maximal amount of dry eye severity symptoms and 0 being the minimal amount or absence of dry eye symptoms.
Change from Baseline to Week 4 in SANDE frequency sub-score (0-100 point VAS) | Baseline to Week 4
  The SANDE frequency sub-score ranges from 0 to 100 with 100 being the maximal amount of dry eye symptoms frequency and 0 being the minimal amount or absence of dry eye symptoms frequency.
Change from Baseline to Week 4 in conjunctival lissamine green staining | Baseline to Week 4
  Lissamine staining is measured by the 0-5 point Oxford grading scale. 0 represents no staining and 5 represents maximal/severe staining and abnormalities to the conjunctiva. Scores from each of the 3 zones as defined by the Oxford grading scale will be evaluated independently.
Change from Baseline to Week 4 in conjunctival injection | Baseline to Week 4
  Conjunctival injection is scored on a 0-2 grading scale. 0 represents no conjunctival injection and 2 represents maximal/severe conjunctival injection and redness of the eye.
Change from Baseline to Week 4 in tear production as measured by the Schirmer's 1 (unanesthetized) tear secretion test | Baseline to Week 4
  The Schirmer strip will be placed into the lower conjunctival sac at the junction of the lateral and middle thirds, avoiding contact with the cornea. The patient will be instructed to close their eyes gently. After 5 minutes have elapsed, the Schirmer test strip will be removed and the length of the tear absorption on the strip will be measured (millimeters/5 minutes).
Change from Baseline to Week 4 in lid margin Vascularity (V) score | Baseline to Week 4
  The lid margin V score is graded on a scale of 0-4 by the vascularization of the lower lid margin between the anterior and posterior edges of the lid. 0 represents absence/minimal vascularization of the lid margin and 4 represents severe/maximal abnormal vascularization.
Change from Baseline to Week 4 in Avascular Zone (Zone A) inflammation score | Baseline to Week 4
  Zone A will be graded on a scale of 0-4 by the hyperemia and vascularization of the normally avascular region of the palpebral conjunctiva ≤1mm posterior to the posterior tarsal edge. 0 represents absence/minimal hyperemia and vascularization and 4 represents severe/maximal abnormal hyperemia and vascularization.
Change from Baseline to Week 4 in Palpebral Conjunctival Redness (PCR) score | Baseline to Week 4
  PCR will be graded by the hyperemia of the palpebral conjunctiva of the lower eyelid on a 0-100 Validated Bulbar Redness (VBR) scale. 0 represents minimal/normal redness and 100 represents maximal/severe redness.

CONTACTS AND LOCATIONS:
Locations (1):
- Richard W Yee, MD PLLC, Bellaire, Texas, United States